CLINICAL TRIAL: NCT01021059
Title: A Phase I Study of Intravenous Recombinant Human IL-15(rhIL-15) in Adults With Metastatic Malignant Melanoma and Metastatic Renal Cell Cancer
Brief Title: A Phase I Study of Intravenous Recombinant Human IL-15 in Adults With Refractory Metastatic Malignant Melanoma and Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100021; 10-C-0021
Record Dates: First submitted 2009-11-25; First posted 2009-11-26 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2016-10-25

CONDITIONS: Melanoma; Carcinoma, Renal Cell
Keywords: Biological Effects of rhIL-15; Estimate Antitumor Activity; rhIL-15 Pharmacokinetics; Dose and Safety Determination of IL-15; Kidney Cancer; Melanoma; Renal Cell Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Kidney Neoplasms

ARMS (1):
- 1 (Experimental): rh IL-15 daily for 12 days of 42 days cycle.
  Interventions: Biological: rh IL-15

INTERVENTIONS:
Biological: rh IL-15 — rh IL-15 daily for 12 days of 42 days cycle. Additional cycles may be given if patient is responding to therapy.

SUMMARY:
Background:

* Recombinant human interleukin-15 (rhIL-15) is a substance that is naturally produced in the body that has many properties that increase the activity and strength of the immune system, the body s natural defense system. It is hoped that rhIL-15 can boost or strengthen patients immune systems and restore immune responses against cancer and infectious diseases like HIV.
* rhIL-15 is being studied in patients with malignant melanoma, an aggressive type of skin cancer, and in patients with renal cell carcinoma, a type of kidney cancer that has spread to other parts of the body. Researchers are interested in determining if rhIL-15 can help stimulate the immune system and aid in the treatment process for cancers that have not responded well to standard therapies.

Objectives:

* To determine whether rhIL-15 is safe and effective in the treatment of metastatic malignant melanoma or metastatic renal cell carcinoma
* To examine how the body processes rhIL-15 after each infusion and determine how it acts on the treated cancer.

Eligibility:

* Patients older than 18 years of age that have been diagnosed with metastatic malignant melanoma or metastatic renal cell carcinoma that has not responded to standard treatments.
* Eligible patients may not have received prior treatment with interleukin-2.

Design:

* Prior to treatment, patients will have baseline blood tests and imaging scans.
* Participants will be admitted to an in-patient unit of the NIH Clinical Center for this treatment. rhIL-15 will be given intravenously once a day for 12 consecutive days, for a total of twelve doses of the drug. The injection of rhIL-15 will take about 30 minutes. Patients will be evaluated daily before each treatment and more frequently if necessary.
* During the 12-day treatment and for at least 42 days from the start of the treatment, patients will be closely followed for possible side effects and for tumor response. Blood will be drawn frequently for monitoring purposes, and other procedures such as chest x-rays and imaging scans will be performed to monitor the state of the tumor and the patient response to treatment.
* After completing the rhIL-15 treatment and discharge from the hospital, patients will have an evaluation with a member of the research team once a week from the end of the treatment period to 42 days from the start of the treatment.
* Study doctors may ask patients to return for evaluation (including blood draws) at 3 and 6 months after the completion of the treatment, checking for potential long-term effects or toxicity of the treatment.

Background:

* Recombinant human interleukin-15 (rhIL-15) is a substance that is naturally produced in the body that has many properties that increase the activity and strength of the immune system, the body s natural defense system. It is hoped that rhIL-15 can boost or strengthen patients immune systems and restore immune responses against cancer and infectious diseases like HIV.
* rhIL-15 is being studied in patients with malignant melanoma, an aggressive type of skin cancer, and in patients with renal cell carcinoma, a type of kidney cancer that has spread to other parts of the body. Researchers are interested in determining if rhIL-15 can help stimulate the immune system and aid in the treatment process for cancers that have not responded well to standard therapies.

Objectives:

* To determine whether rhIL-15 is safe and effective in the treatment of metastatic malignant melanoma or metastatic renal cell carcinoma
* To examine how the body processes rhIL-15 after each infusion and determine how it acts on the treated cancer.

Eligibility:

* Patients older than 18 years of age that have been diagnosed with metastatic malignant melanoma or metastatic renal cell carcinoma that has not responded to standard treatments.
* Eligible patients may not have received prior treatment with interleukin-2.

Design:

* Prior to treatment, patients will have baseline blood tests and imaging scans.
* Participants will be admitted to an in-patient unit of the NIH Clinical Center for this treatment. rhIL-15 will be given intravenously once a day for 12 consecutive days, for a total of twelve doses of the drug. The injection of rhIL-15 will take about 30 minutes. Patients will be evaluated daily before each treatment and more frequently if necessary.
* During the 12-day treatment and for at least 42 days from the start of the treatment, patients will be closely followed for possible side effects and for tumor response. Blood will be drawn frequently for monitoring purposes, and other procedures such as chest x-rays and imaging scans will be performed to monitor the state of the tumor and the patient response to treatment.
* After completi...

DETAILED DESCRIPTION:
Background:

* Interleukin-15 (IL-15) is a powerful immunostimulatory cytokine with a broad range of biological activities.
* In contrast to IL-2, IL-15 inhibits the activation-induced cell death (AICD) of T-cells and is not involved in the maintenance of CD4+CD25+ T regulatory cells that act as inhibitory checkpoints on the immune response.
* IL-15 is involved in the proliferation, differentiation and activation of CD8+ T-cells and NK-cells, and the maintenance of long term CD8+ memory T-cells.
* In preclinical studies, vaccinia-based vaccines expressing IL-15 induced long lasting, high-avidity cytotoxic CD8+ T-lymphocyte (CTL) mediated immunity, whereas the immunity mediated by IL-2 expressing vaccines was short-lived. Furthermore, IL-15 can overcome the lack of CD4 help in CTL induction.
* IL-15 is highly active against a number of syngeneic mouse tumor models and it is also effective in augmenting the activity of NK-cells and CD8+ T-cells in rhesus macaques indicating that it may be active against human cancers.

Objectives:

* The primary objective of this trial is to determine the safety, toxicity profile, dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of intravenous recombinant human IL-15 (rhIL-15) administered as a daily intravenous bolus infusion for 12 consecutive days in subjects with metastatic malignant melanoma and renal cell cancer.
* Secondary objectives include determination of rhIL-15 pharmacokinetics, in particular the time course of the decline of rhIL-15 from the serum following intravenous administration and the definition of the immunogenicity of rhIL-15 in subjects receiving this drug.
* To characterize the biological effects of rhIL-15 on the proportions and absolute numbers of circulating NK-cells, and CD45RO+CD8+ T-cells and central or effector memory subsets based on expression of CD28, CD95, CCR7 and CD62L by flow cytometry and to determine its effects on the plasma levels of pro-inflammatory cytokines.
* Obtain preliminary information on the antitumor effects of repeat cycles of rhIL-15 in patients with metastatic malignant melanoma and renal cell cancer.

Eligibility Criteria:

* Patients greater than or equal to 18 years-old with pathologically confirmed metastatic malignant melanoma or metastatic renal cell cancer.
* Patients with metastatic renal cell cancer must either have refused treatment with, failed to tolerate, or have progressive disease after receiving sorafenib or sunitinib, and temsirolimus.
* Patients with measurable disease.
* Absolute granulocyte count (AGC) of at least 1500/mm(3) and a platelet count of at least 75,000/mm(3).

Design:

* This is a single institution, open-label, non-randomized 3 + 3 design phase I dose-escalation study to determine the safety, toxicity and MTD of rhIL-15 in patients with metastatic malignant melanoma and renal cell cancer.
* Groups of 3 to 6 patients will receive rhIL-15 at doses of 0.3, 1, 3, 7, 10, 15, 20 or 25 mcg/kg/day for 12 days provided that DLT had not been observed.
* Correlative protocol studies will be obtained prior to treatment and at specific times points during and after treatment including pharmacokinetics for the clearance of rhIL-15 from the serum, immunogenicity testing for the development of neutralizing anti-rhIL-15 antibodies and immunological study endpoint evaluation for the effect of rhIL-15 on immune cell subset populations and pro-inflammatory cytokine levels in the peripheral blood.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years.
* Diagnosis of metastatic malignant melanoma or metastatic renal cell cancer confirmed by the Laboratory of Pathology, NCI.
* Patients must have metastatic malignant melanoma or metastatic renal cell cancer (AJCC stage IV [M1] or equivalent disease). Metastatic renal cell cancer patients must either have refused treatment with, have been unable to tolerate or have experienced progressive disease after treatment with sorafenib or sunitinib, and temsirolimus.
* Patients must have measurable disease.
* DLCO/VA and FEV-1.0 greater than 50% of predicted on pulmonary function tests.
* AST and ALT less than 3 times the upper limit of normal.
* Absolute neutrophil count greater than or equal to 1,500/mm(3).
* Platelets greater than or equal to 75,000/mm(3).
* PT/PTT within 1.5 times upper limit of normal. Patients with a history of DVT and who are on anticoagulation therapy may be eligible, provided their DVT was at least 8 weeks prior to enrollment and they have had no further complications.
* Karnofsky performance status greater than or equal to 70% (ECOG less than or equal to 1)
* Serum creatinine of less than or equal to 1.5 times the upper limit of normal.
* CNS metastases: Patients who remain asymptomatic after successful definitive treatment of brain metastases (i.e., surgical resection, curative whole brain irradiation, stereotactic radiation therapy, or a combination of these) demonstrating stable or improved radiographic appearance on MRI scan greater than or equal to 3 months after completion of treatment and no signs of cerebral edema are eligible.

EXCLUSION CRITERIA:

* Patients must not have received any systemic corticosteroid therapy for 3 weeks prior to the start of therapy with the exception of physiological replacement doses of cortisone acetate or equivalent.
* Patients must not have received any cytotoxic therapy, immunotherapy, antitumor vaccines or monoclonal antibodies in the 4 weeks prior to the start of the study.
* History of any hematopoietic malignancy.
* Life expectancy of less than 3 months.
* Presence of serum antibodies to IL-15.
* Patients must not have a marked baseline prolongation of QT/QTc interval (e.g., demonstration of a QTc interval greater than 500 milliseconds (ms)).
* Documented HIV, active or chronic hepatitis B, hepatitis C or HTLV-I infection.

  * A positive hepatitis B serology indicative of previous immunization (i.e., HBsAb positive and HBc Ab negative), or a fully resolved acute HBV infection is not an exclusion criterion.
  * A positive hepatitis C serology is an exclusion criterion.
* Concurrent anticancer therapy (Including other investigational agents).
* History of severe asthma, presently on chronic medications (a history of mild asthma not requiring therapy is eligible).
* History of autoimmune disease, with the exception of an autoimmune event associated with prior ipilimumab (anti-CTLA-4) therapy that has completely resolved for a period of more than 4 weeks.
* Inability or refusal to practice effective contraception during therapy or the presence of pregnancy or active breastfeeding (Men and women of childbearing potential must use an effective method of birth control or abstinence during treatment and for four months after completion of treatment).
* History of medical or psychiatric disease, active substance abuse or social circumstances which in the view of the Principal Investigator, would preclude safe treatment.
* Patients with cognitive impairment or likely to develop cognitive impairment while on study.
* Inability to give informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-11-10; Primary Completion 2013-05-31 (Actual); Study Completion 2016-10-25 (Actual)

PRIMARY OUTCOMES:
Determine the safety, toxicity profile, dose-limiting toxicity and a maximum tolerated dose if IV recombinant Human IL-15 administered in melanoma and renal cell cancers. | After first cycle

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Waldmann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Waldmann TA, Tagaya Y. The multifaceted regulation of interleukin-15 expression and the role of this cytokine in NK cell differentiation and host response to intracellular pathogens. Annu Rev Immunol. 1999;17:19-49. doi: 10.1146/annurev.immunol.17.1.19. PMID 10358752
- [Background] Waldmann TA, Dubois S, Tagaya Y. Contrasting roles of IL-2 and IL-15 in the life and death of lymphocytes: implications for immunotherapy. Immunity. 2001 Feb;14(2):105-10. No abstract available. PMID 11239443
- [Background] Waldmann TA. The biology of interleukin-2 and interleukin-15: implications for cancer therapy and vaccine design. Nat Rev Immunol. 2006 Aug;6(8):595-601. doi: 10.1038/nri1901. PMID 16868550
- [Derived] Conlon KC, Lugli E, Welles HC, Rosenberg SA, Fojo AT, Morris JC, Fleisher TA, Dubois SP, Perera LP, Stewart DM, Goldman CK, Bryant BR, Decker JM, Chen J, Worthy TA, Figg WD Sr, Peer CJ, Sneller MC, Lane HC, Yovandich JL, Creekmore SP, Roederer M, Waldmann TA. Redistribution, hyperproliferation, activation of natural killer cells and CD8 T cells, and cytokine production during first-in-human clinical trial of recombinant human interleukin-15 in patients with cancer. J Clin Oncol. 2015 Jan 1;33(1):74-82. doi: 10.1200/JCO.2014.57.3329. Epub 2014 Nov 17. PMID 25403209